CLINICAL TRIAL: NCT05171231
Title: Observational, Multicenter, Prospective Clinical Study, Measuring the Performance and Safety of the Surgical Hemostatic Agent "HEMOCOLLAGENE®" in Patients Requiring Oral Surgery
Brief Title: Performance and Safety of the Surgical Hemostatic Agent "HEMOCOLLAGENE®" in Patients Requiring Oral Surgery
Status: Completed | Type: Observational
Sponsor: Septodont (Industry)
Collaborators: Symatese (Industry); Recherche Clinique en Odontologie (ReCOL) (Network); EndoData (Unknown)
Responsible Party: Sponsor
Other Study IDs: HEM 2021-07; 2021-A01764-37 (Registry Identifier: French ID-RCB)
Record Dates: First submitted 2021-11-22; First posted 2021-12-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Oral Hemorrhage
Keywords: Surgical Hemostatic; Oral Surgery
MeSH Terms: conditions — Oral Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: HEMOCOLLAGENE® : Sterile absorbable hemostatic sponges based on bovine collagen - class III MD — HEMOCOLLAGENE® is an absorbable, sterile and hemostatic sponge, composed of type I undenatured, native and lyophilized bovine collagen (0.027 g per sponge).
  HEMOCOLLAGENE® will be inserted into oral sites (mainly the alveoli dental) after post-extraction or post-invasive dental surgical procedure, in case of bleeding not controled by usual hemostatic method. HEMOCOLLAGENE® will be let in place and will undergo a complete and natural absorption after several weeks.

SUMMARY:
The aim of this study is to collect performance and safety data relating to the use and the follow-up of the HEMOCOLLAGENE® medical device in routine clinical practice from various hospitals and medical centers in oral dental surgery.

Patients will The data collected from the Post-Market Clinical Follow-up study will be used to support the regulatory requirements of post-market monitoring (risk management, residual risks, instructions for use...) and to increase the manufacturer's clinical data. Patients will be followed for 1 month.

Adverse events (safety) and device performance will be collected by the dentist during the routine follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring oral surgery
* Patient with a bleeding requiring the use of an adjuvant hemostatic
* Patient implanted with HEMOCOLLAGENE® in dental surgery.
* Patient who signed his informed consent form

Exclusion Criteria:

* Inform Consent not signed
* Patients with acute oral infection.
* Patients with an unstable hemodynamic state (acute and/or chronic cardiovascular pathology, low arterial pressure, cardiac rhythm problem)
* Pregnant and / or breastfeeding patients.
* Patient with hypersensitivity or allergy to bovine collagen

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is made with the recruitment of participating centers which included at least one patient.
  The analysis will be carried out on the patients included with evaluable observation sheets . The evaluability of a form will be defined during the development of the analysis plan according to the number of missing data and the nature of missing data.
  The analysis sets are defined below:
  * Intented-to-treat (ITT) population: The ITT population consists of all subjects not opposed to the use of their clinical data and implanted by the HEMOCOLLAGENE® medical device. This population will be the primary population analysis for safety and efficacy.
  * Per Protocol (PP): The PP population includes all the patients implanted by the medical device HEMOCOLLAGENE® without any major deviation from the protocol. Protocol violations will be graded (major / minor) when reviewing data before database lock. This population will be the secondary population analysis.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Hemostatic Performance at 5 minutes | 5 minutes after treatment onset
  Evaluation of the stop of the bleeding 5 minutes after using HEMOCOLLAGENE®.

SECONDARY OUTCOMES:
Rate of overall adverse events | From treatment onset to 30 days
  overall Safety assessment
Rate of device related adverse events | From treatment onset to 30 days
  Safety assessment relating to the medical device
Wound Healing | At 30 days
  Evaluation of the wound healing using the Landry Score (from "1 - Very Poor" to "5 - Excellent")
Ease of the use of Hemocollagene by the Dentist | At day 0, after using the treatment
  Satisfaction of the dentist on the use and the quality of HEMOCOLLAGENE® :
  * Data relating to the hemostatic agent HEMOCOLLAGENE® (number, reference, quality before and during use).
  * The technique for using HEMOCOLLAGENE® (cutting before or after application, removal or not for hemostasis, fixing).
  * The intraoperative satisfaction of the practitioner.
Rate of hemostatic time at 10 minutes in case persistant bleeding | 10 minutes after treatment onset
  Percentage of patients with a bleeding stopped 10 minutes after treatment onset in case of persistant bleeding
Rate of persistant bleeding | 5 minutes after treatment onset
  Percentage of patients with a bleeding not stopped 5 minutes after treatment onset

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Grosgogeat, MD, PhD, Study Director — CHU de Lyon, France
Locations (10):
- Belgium (2):
  - Cabinet Dento Médical, cabinet de Nivelles, Baulers
  - Cabinet Dentaire, Brussels
- France (8):
  - Cabinet dentaire, Chassieu
  - SCM Chirurgie Dentaire Opéra, Lyon
  - Cabinet Medical, Lyon
  - HCL-Hospices Civil de Lyon, Lyon
  - Cabinet dentaire Grange-Blanche, Lyon
  - APHP- Hôpital de la Pitié Salpetrière, Paris
  - Cabinet dentaire, Roanne
  - Cabinet dentaire, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guillet, Marie, et al. "Adjuvant Hemostasis in Dental Surgery: Real-Life Practice Data in The Observational, Multi-Center, Prospective, Hemocollagene Clinical Trial." International Journal of Health & Medical Research 3.12 (2024).